CLINICAL TRIAL: NCT05290233
Title: Time Restricted Eating Plus Exercise for Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kelsey Nicole Dipman Gabel, Clinical Assistant Professor and Postdoctoral Researcher, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0279
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Intermittent Fasting; Pre Diabetes; Cognitive Decline
MeSH Terms: conditions — Intermittent Fasting; Glucose Intolerance; Cognitive Dysfunction | interventions — Trehalase; Exercise

STUDY DESIGN:
Intervention Model Description: A 12-week randomized, parallel-arm pilot trial will compare the effects of 1) TRE combined with resistance training (TRE-RT) to 2) TRE combined with aerobic training (TRE-AT) in older adults with overweight or obesity and pre-diabetes
Who Masked: Outcomes Assessor
Masking Description: blood sample analysis will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRE+RT (Experimental): Participants will confine eating between either 10am-6pm or 12-8pm and fast from 6pm-10am or 8pm-12pm daily combined with 3-4 days of supervised resistance training per week.
  Interventions: Behavioral: TRE + Exercise
- TRE+AT (Active Comparator): Participants will confine eating between either 10am-6pm or 12-8pm and fast from 6pm-10am or 8pm-12pm daily combined with 3-4 days of supervised aerobic training per week.
  Interventions: Behavioral: TRE + Exercise

INTERVENTIONS:
Behavioral: TRE + Exercise — We will compare the effects of TRE combined with resistance exercise versus TRE combined with aerobic training.
  Other Names:
  resistance training endurance exercise

SUMMARY:
Time restricted eating (TRE) is currently the most popular form of intermittent fasting which involves confining the eating window to 8-10 hours (h) and fasting for the remaining hours of the day. TRE is unique in that during the eating window, individuals are not required to count calories or monitor food intake in any way, resulting in high adherence. Accumulating evidence suggests that TRE produces a natural energy deficit of ~350-500 kcal/d. Physical activity in combination with a healthy diet pattern is recommended for older adults. While aerobic type exercise is the most commonly recommended, retention of lean mass via resistance training, especially in older adults, may be more effective at improving mobility, neurological and psychological function, executive and cognitive functioning, and processing speed. TRE combined with physical activity has not been examined in older adults or in people with overweight or obesity. This study holds the potential to 1) decrease body weight 2) improve lean mass 3) improve insulin sensitivity, and 4) improve attention, executive functioning, and processing speed in older adults. The aims of this study will examine the effect of TRE combined with either resistance training or aerobic training on body weight, body composition, metabolic disease risk, and cognition in adults over age 50. It is hypothesized that the TRE combined with resistance training group will see the most significant improvements in body composition, insulin sensitivity and cognition due to lean mass accretion.

DETAILED DESCRIPTION:
Time restricted eating (TRE) is currently the most popular form of intermittent fasting which involves confining the eating window to 8-10 hours (h) and fasting for the remaining hours of the day. TRE is unique in that during the eating window, individuals are not required to count calories or monitor food intake in any way, resulting in high adherence. Accumulating evidence suggests that TRE produces a natural energy deficit of ~350-500 kcal/d. Physical activity in combination with a healthy diet pattern is recommended for older adults. While aerobic type exercise is the most commonly recommended, retention of lean mass via resistance training, especially in older adults, may be more effective at improving mobility, neurological and psychological function, executive and cognitive functioning, and processing speed. T TRE combined with physical activity has not been examined in older adults or in people with overweight or obesity. This study holds the potential to 1) decrease body weight 2) improve lean mass 3) improve insulin sensitivity, and 4) improve attention, executive functioning, and processing speed in older adults. This study will examine the effect of TRE combined with either resistance training or aerobic training on body weight, body composition, metabolic disease risk, and cognition in adults over age 50. It is hypothesized that the TRE combined with resistance training group will see the most significant improvements in body composition, insulin sensitivity and cognition due to lean mass accretion.

ELIGIBILITY:
Inclusion Criteria:

* Adults with obesity (BMI between 30-50kg/m2)
* pre-diabetes (fasting glucose: 100-125 mg/dl or HBA1c 5.7%-6.4% or OGTT ≥ 200 mg/dl)
* sedentary or lightly active (<7,500 steps/day)
* between the ages of 50-80 years

Exclusion Criteria:

* diagnosed with T1DM or T2DM (fasting glucose: >126 mg/dl, 2-h glucose OGTT ≥ 200 mg/dl,
* HbA1c: >6.5%)
* Individuals with a history of eating disorders
* shift workers
* Individuals taking drugs to control body weight and glucose (including metformin)
* individuals who are not weight stable (weight gain or loss > 4 kg) 3 months prior to the intervention
* mobility disorders or individuals unable to exercise for 40-60 minutes 3-4 days/week
* Individuals diagnosed with comorbidities impacting cognition, including major/mild neurocognitive disorder, cerebrovascular disease (e.g., stroke, aneurysm, arteriovenous malformation), traumatic brain injury, epilepsy, or major psychiatric disorder (e.g., schizophrenia, bipolar disorder, substance use disorder)
* Individuals who are unable to adequately report dietary intake or physical activity
* Smokers

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Lean mass | change from week 1 to week 12
  fat free mass will be measured via DXA

SECONDARY OUTCOMES:
body weight | change kg of body weight from week 1 to week 12
  Body weight assessed to the nearest 0.25 kg every week without shoes and in light clothing using a balance beam scale (HealthOMeter, Boca Raton, FL).
fat mass | change kg of body weight from week 1 to week 12
  fat mass will be measured via DXA
Visceral fat mass | change kg of body weight from week 1 to week 12
  visceral fat mass will be measured via DXA
Insulin | change from week 1 to week 12
  measured by enzymatic kit (uIU/ml)^4
glucose | change from week 1 to week 12
  measured by enzymatic kit (mg/dl)
HbA1c | change from week 1 to week 12
  measured by enzymatic kit (mmol/mol)
Attention | Change from week 1 to week 12
  National Institutes of Health Toolbox Cognition Battery
executive function | Change from week 1 to week 12
  National Institutes of Health Toolbox Cognition Battery
processing speed | Change from week 1 to week 12
  National Institutes of Health Toolbox Cognition Battery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No